CLINICAL TRIAL: NCT03044509
Title: Evaluation and Validation of Novel Immunodiagnostic Tests for Childhood Tuberculosis Infection and Disease in Switzerland. The CITRUS (ChIldhood TubeRcUlosis in Switzerland) Study.
Brief Title: Diagnosis of Tuberculosis in Swiss Children
Acronym: CITRUS
Status: Recruiting | Type: Observational
Sponsor: University Children's Hospital Basel (Other)
Collaborators: Ospedale Regionale Bellinzona e Valli (Other); Insel Gruppe AG, University Hospital Bern (Other); University of Lausanne Hospitals (Other); University Hospital, Geneva (Other); Luzerner Kantonsspital (Other); Cantonal Hospital of St. Gallen (Other); University Children's Hospital, Zurich (Other); Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, Dr. Nicole Ritz, MD/PhD, PI, University Children's Hospital Basel
Other Study IDs: CITRUS
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Tuberculosis; Mycobacterium Tuberculosis
Keywords: Immunodiagnostics tests; TB exposure; Latent TB; TB disease; Biomarkers; Metabolomics; NMR
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples Without DNA — For each child a total blood volume of 7.5 ml will be required for this study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- TB exposure
  Interventions: Diagnostic Test: Secreted cytokine assay; Diagnostic Test: Intracellular cytokine assay
- TB infection (latent TB)
  Interventions: Diagnostic Test: Secreted cytokine assay; Diagnostic Test: Intracellular cytokine assay
- TB disease (active TB)
  Interventions: Diagnostic Test: Secreted cytokine assay; Diagnostic Test: Intracellular cytokine assay

INTERVENTIONS:
Diagnostic Test: Secreted cytokine assay — Blood collected in a sodium-heparin tube will be used for the assay using novel TB-specific antigens. After incubation the supernatant will be harvested and cryopreserved at -80 °C for further testing of cytokines. Cytokines will be measured using a bead-based multiplex assay reader (MAGPIX, Luminex Crop., Austin, USA).
Diagnostic Test: Intracellular cytokine assay — Blood will be stimulated with recombinant MTB-specific antigens, ESAT-6, CFP-10, positive control or left unstimulated. Following an initial duration of stimulation, Brefeldin-A will be added and the blood incubated for a further 5 hours. White cells will be fixed and cryopreserved at - 80°. Batched analysis within 6 months of cryopreservation will be done using multi-colour flow cytometry.

SUMMARY:
1. The primary objective is to improve the sensitivity of novel immunodiagnostic tests for detection of TB disease in children.
2. The secondary objective is to determine biomarkers that discriminate children with TB infection and disease.

DETAILED DESCRIPTION:
1. This will be done by measuring a variety of parameters in the blood samples and compare them with the current diagnostic gold standard for TB or for culture/NAAT non-confirmed TB cases a consensus case definition is used.

   Currently available immunodiagnostic tests (IGRA/TST) will be compared to novel immunodiagnostic tests which will include:
   * several novel, additional M. tuberculosis-specific Antigens
   * cytokines that are highly expressed
2. Since there is no diagnostic gold standard for TB infection we will rely on a clinical composite reference standard for diagnosing TB infection. Biomarkers will be determined by:

   * including M. tuberculosis-specific antigens that are specifically expressed in either TB infection or disease,
   * measuring phenotypes and cytokine production of M. tuberculosis-specific cells.
   * performing NMR Analysis with biofluids in order to identify metabolomic signatures in patients with TB disease and TB infection

ELIGIBILITY:
Inclusion Criteria:

* all children / adolescents < 18 years of age undergoing evaluation for TB exposure, infection or disease.

Exclusion Criteria:

* children / adolescents with TB infection or disease who have already been started on anti-mycobacterial treatment, children who have been treated for TB previously.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: It will be a national multicentre study in Switzerland. Children will be recruited within SwissPedNet, the Swiss Research Network of Clinical Paediatric Hubs, which includes five University Children's Hospitals (Basel, Bern, Geneva, Lausanne and Zürich) and four cantonal A-clinics (Aarau, Bellinzona, Luzern and St. Gallen). Currently approximately 20-30 children with TB disease are notified in Switzerland each year. For TB infection in children there are no data available in Switzerland. However, data from the "Lungenliga Schweiz" show that in 2014, at least 232 children were examined for a TB contact investigation (correspondence with Jean-Pierre Zellweger and Jean-Marie Egger, Lungenliga Schweiz 13.08.2015). Of these 13 % (i.e. around 30 children) are categorized as TB infection per year.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2017-05-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of immunodiagnostic tests for TB in children. | 27 months
  Based on current evidence it is estimated that the sensitivity of the immunodiagnostic tests with regard to the identification of patients with TB infection or disease versus no TB is approximately 80 %. By applying a sample size approximation a minimum sample size of 126 patients with TB infection or disease (with a precision given by a 95 % confidence interval with a width of 20 %) will be needed to statistically show a significant result.

SECONDARY OUTCOMES:
Indicative markers identification for TB infection and disease distinction | 27 months
  A minimum sample size of 84 patients with TB infection is needed (with a precision given by a 95 % confidence interval with a width of 30 %). Among patients with TB infection or TB disease, a novel test is used to discriminate between these patient groups. It is estimated that the sensitivity of this test with regard to the identification of patients with TB infection (secondary outcome) is approximately 60 %.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Ritz, Prof Dr med, Principal Investigator — UKBB
Locations (8):
- Switzerland (8):
  - Kantonspital Aarau, Aarau
  - Nina Vaezipour, Basel
  - Ospedale Regionale di Bellinzona, Bellinzona
  - Inselspital Bern, Bern
  - Hôpital des enfants - HUG, Geneva
  - Kinserspital Luzern, Lucerne
  - Kinderspital St Gallen, Sankt Gallen
  - Kinderklinik Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neudecker D, Fritschi N, Sutter T, Lu LL, Lu P, Tebruegge M, Santiago-Garcia B, Ritz N. Evaluation of serological assays for the diagnosis of childhood tuberculosis disease: a study protocol. BMC Infect Dis. 2024 May 10;24(1):481. doi: 10.1186/s12879-024-09359-0. PMID 38730343